CLINICAL TRIAL: NCT00449345
Title: Screening for Latent Tuberculosis in Healthcare Workers With Quantiferon-Gold Assay: A Cost-Effectiveness Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Other Study IDs: 2006055
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Latent Tuberculosis Infection
Keywords: Latent tuberculosis infection; Health care workers; Tuberculin skin test; Mantoux skin test; Interferon gamma; Quantiferon; Cost effectiveness
MeSH Terms: conditions — Latent Tuberculosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood test for Quantiferon-GOLD assay

SUMMARY:
The ministry of health in Israel requires all health-care workers to undergo screening for latent Tuberculosis infection (LTBI) prior to starting work. This is based on the Mantoux skin test, which is notoriously unreliable.

In recent years, more specific and sensitive tests based on interferon-gamma secretion to TB antigens have come to market, and most current evidence shows that many mantoux positive persons do not have LTBI. Quantiferon-GOLD is one of these assays.

In this prospective study, we will draw blood for the Quantiferon-GOLD assay in parallel to conventional testing, and perform a cost-effectiveness analysis of the cost of the investigation and treatment of LTBI in health-care workers.

We hypothesize that in spite of the cost of screening healthcare workers with Quantiferon-GOLD tests, the reduction in need for LTBI treatment and associated costs will render the test cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Health care worker undergoing screening for LTBI

Exclusion Criteria:

* Previous tuberculosis or treatment for LTBI
* Immunosuppressed due to drug treatment, HIV, organ transplant
* Recent TB contacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Community Tuberculosis service, Rehovot, Israel